CLINICAL TRIAL: NCT00428428
Title: Pharmacological Modulation of the Intrarenal Pressure During Endourological Procedures in the Upper Urinary Tract
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Fredericia Hosptial (Other)
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: HJ2; EudraCT nummer: 2006-005756-32
Record Dates: First submitted 2007-01-29; First posted 2007-01-30 (Estimated); Last update posted 2007-11-16 (Estimated); Status verified 2007-11

CONDITIONS: Kidney Stone; Unexplained Haematuria; Benignant Tumour Mass in the Upper Urinary Tract
Keywords: kidney stone; ureteroscopy
MeSH Terms: conditions — Kidney Calculi | interventions — Isoproterenol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Placebo Comparator): Saline irrigation
  Interventions: Drug: Isoproterenol
- 2 (Active Comparator): ISO irrigation
  Interventions: Drug: Isoproterenol

INTERVENTIONS:
Drug: Isoproterenol — ISO 0.1 microgram/ml, 8 ml/min irrigation compared to saline irrigation

SUMMARY:
The purpose of the study is to examine the effect of endoluminally administrated isoproterenol on pelvic pressure increase during flexible ureterorenoscopy in 14 humans. We propose that isoproterenol has potential of reducing intrarenal pressure during ureterorenoscopies. Lower intrarenal pressures may have the advantage of facilitating the procedure and reducing intraoperative complications as bleeding and infections.

ELIGIBILITY:
Inclusion Criteria:

* Indication for ureterorenoscopy
* Age> 18 years
* Normal blood pressure

Exclusion Criteria:

* Malignant disease in the upper urinary tract
* Heart disease
* Allergy to Isoproterenol
* Use of α-blocking or β-blocking medicine
* Use of Calcium-antagonists
* Use of NSAIDs the last 48 hours
* Present stone or JJ-stent in the ureter
* Neurologic disease in the bladder
* Pregnancy
* Nursing mothers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2007-02; Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
pelvic pressure

CONTACTS AND LOCATIONS:
Overall Officials: Palle JS Osther, PhD, MD, Study Director — Dp. of Urology, Fredericia & Kolding Hospitals, Fredericia, denmark
Locations (1):
- Dp. of Urology, Fredericia & Kolding Hospitals, Fredericia, Fredericia, Denmark